CLINICAL TRIAL: NCT06367946
Title: Mechanism Study Under the Role of Tissue Kallikrein-related Peptidase 8 (KLK8)-Induced Senescence of Pulmonary Vascular Endothelial Cells in Ventilator-induced Lung Injury in Elderly People.
Brief Title: Mechanism Study of Ventilator-Induced Lung Injury in Elderly People.
Status: Recruiting | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Lai Jiang, 021-25077820, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XH-24-0093
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Ventilator-Induced Lung Injury
MeSH Terms: conditions — Ventilator-Induced Lung Injury | interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. Lung tissues from patients undergoing partial lung resection surgery
  2. Peripheral blood from patients undergoing general anesthesia surgery with mechanical ventilation before mechanical ventilation and after mechanical ventilation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Under 40 years old: Patients undergoing surgery with mechanical ventilation who are under 40 years old
  Interventions: Procedure: mechanical ventilation
- 40-50 years old: Patients undergoing surgery with mechanical ventilation who are 40-50 years old
  Interventions: Procedure: mechanical ventilation
- 50-60 years old: Patients undergoing surgery with mechanical ventilation who are 50-60 years old
  Interventions: Procedure: mechanical ventilation
- 60-70 years old: Patients undergoing surgery with mechanical ventilation who are 60-70 years old
  Interventions: Procedure: mechanical ventilation
- 70-80 years old: Patients undergoing surgery with mechanical ventilation who are 70-80 years old
  Interventions: Procedure: mechanical ventilation
- Over 80 years old: Patients undergoing surgery with mechanical ventilation who are over 80 years old
  Interventions: Procedure: mechanical ventilation

INTERVENTIONS:
Procedure: mechanical ventilation — Mechanical ventilation is machine-delivered flow of gases to both oxygenate and ventilate a patient who is unable to maintain physiological gas exchange.

SUMMARY:
1. We collect lung tissues from patients with different ages and confirm that KLK8 expression is positively correlated with age.
2. We collect peripheral blood from patients with different ages and duration of mechanical ventilation to explore the correlation between the degree of endothelial/epithelial damage, age and duration of mechanical ventilation.

DETAILED DESCRIPTION:
1. We collect lung tissues from patients with different ages and confirm that KLK8 expression is positively correlated with age. All clinical samples have been collected and tested uniformly. Correlation analysis between KLK8 and age will be performed by using Statistical Package for the Social Sciences (SPSS) 22.0 software, and P<0.05 indicates a statistically significant difference. The obtained clinical data should be recorded on survey forms, and researchers should verify patient information by recording basic information such as age and gender.
2. We collect peripheral blood from patients with different ages and duration of mechanical ventilation to explore the correlation between the degree of endothelial/epithelial damage, age and duration of mechanical ventilation. All clinical samples have been collected and tested uniformly. Correlation analysis between endothelial/epithelial damage index, age and duration of mechanical ventilation will be performed by using SPSS 22.0 software, and P<0.05 indicates a statistically significant difference. The obtained clinical data should be recorded on survey forms, and researchers should verify patient information by recording basic information such as age and gender.

ELIGIBILITY:
Inclusion Criteria:

1. Lung tissues from patients with different ages:

   Patients undergoing elective general anesthesia surgery; Patients undergoing partial lung resection with mechanical ventilation; American Society of Anesthesiology (ASA) grade 2-3;
2. Peripheral blood from patients with different ages and duration of mechanical ventilation:

Patients undergoing elective general anesthesia surgery with mechanical ventilation; ASA grade 2-3;

Exclusion Criteria:

1. Lung tissues from patients with different ages:

   Patients with chronic lung diseases (asthma, chronic obstructive pulmonary disease (COPD), pulmonary heart disease, etc.); Patients with human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), hepatitis D virus (HDV), or receiving immunotherapy; Patients who have recently suffered from pneumonia; Recent history of mechanical ventilation; Patients with thrombotic diseases; Children and pregnant women.
2. Peripheral blood from patients with different ages and duration of mechanical ventilation:

Patients with chronic lung diseases (asthma, COPD, pulmonary heart disease, etc.); Smoking patients; Patients with hypertension/diabetes/coronary heart disease; Patients with HIV, HBV, HCV, HDV, or receiving immunotherapy; Patients who have recently suffered from pneumonia; Recent history of mechanical ventilation; Patients with thrombotic diseases; Children and pregnant women.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We started collecting lung tissues and peripheral blood from patients with mechanical ventilation from June 2023. All clinical samples have been collected and tested uniformly. Correlation analysis between KLK8 and age using SPSS 22.0 software will be performed, and P<0.05 indicates a statistically significant difference. The obtained clinical data should be recorded on survey forms, and researchers should verify patient information by recording basic information such as age and gender.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
KLK8 concentration of lung tissue | 2023.7.1-2024.7.1
  The concentration of KLK8 in lung tissue is determined by ELISA.
Endothelial/epithelial damage index concentration in peripheral blood | 2024.5.1-2024.8.1
  The concentration of endothelial/epithelial damage index in lung tissue is determined by ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Lai Jiang, PhD, Principal Investigator — Department of Anesthesia, Shanghai Xinhua hospital, Shanghai China
Locations (1):
- Shanghai Xinhua hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No